CLINICAL TRIAL: NCT06897579
Title: A Randomized Controlled, Open-label, Multicenter Clinical Trial Evaluating the Efficacy and Safety of Carboplatin/Cisplatin + Etoposide + Bemarituzumab Followed by Bemarituzumab Combined With Anlotinib Versus Carboplatin/Cisplatin + Etoposide + Tislelizumab Followed by Tislelizumab as First-line Treatment for Extensive-stage Small Cell Lung Cancer
Brief Title: Carboplatin/Cisplatin + Etoposide + Benmelstobart Sequential Benmelstobart Combined With Anlotinib Versus Carboplatin/Cisplatin + Etoposide + Tislelizumab Sequential Tislelizumab in the Treatment of Extensive Stage Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TQB2450-ALTN-II-03
Record Dates: First submitted 2025-03-19; First posted 2025-03-27 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2024-11

CONDITIONS: Extensive Stage Small Cell Lung Cancer
MeSH Terms: interventions — Carboplatin; Injections; Cisplatin; Etoposide; tislelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carboplatin/cisplatin + etoposide + benmelstobart + Anlotinib hydrochloride (Experimental): Induction treatment period：Carboplatin for injection/Cisplatin for injection + etoposide injection + benmelstobart injection, intravenous infusion, 21 days 1 cycle (etoposide injection on the 2nd and 3rd day of each cycle) Maintenance treatment period: benmelstobart injection, intravenous drip, 21 days 1 cycle；Anlotinib hydrochloride capsules were taken orally on an empty stomach for 2 consecutive weeks and stopped for 1 week.
  Interventions: Drug: Carboplatin for injection/cisplatin for injection + etoposide injection + benmelstobart injection + Anlotinib hydrochloride capsule
- Carboplatin /Cisplatin + etoposide + Tislelizumab (Active Comparator): Induction treatment period：Carboplatin for injection/Cisplatin for injection + etoposide injection + Tislelizumab injection, intravenous infusion, 21 days, 1 cycle (etoposide injection on the 2nd and 3rd day of each cycle) Maintenance treatment period：Tislelizumab injection, intravenous drip, 21 days 1 cycle.
  Interventions: Drug: Carboplatin for injection/Cisplatin for injection + etoposide injection + Tislelizumab injection

INTERVENTIONS:
Drug: Carboplatin for injection/cisplatin for injection + etoposide injection + benmelstobart injection + Anlotinib hydrochloride capsule — Carboplatin for injection inhibits DNA synthesis, thereby preventing cancer cell division and reproduction/Cisplatin for injection binds to DNA, interfering with DNA replication and transcription processes, Thus inhibiting tumor cell proliferation/etoposide injection interferes with the division process of cancer cells to inhibit their growth and spread/Bemosubebezumab injection is a humanized recombinant anti-Programmed cell death ligand 1 (PD-L1) monoclonal antibody/Anlotinib hydrochloride capsule is a tyrosine kinase inhibitor.
  Arms: Carboplatin/cisplatin + etoposide + benmelstobart + Anlotinib hydrochloride
Drug: Carboplatin for injection/Cisplatin for injection + etoposide injection + Tislelizumab injection — Carboplatin for injection inhibits DNA synthesis and thus prevents the division and reproduction of cancer cells/Cisplatin for injection binds to DNA and interferes with the DNA replication and transcription process, thereby inhibiting the proliferation of tumor cells/etoposide injection interferes with the division process of cancer cells to inhibit their growth and spread/Tislelizumab injection is a humanized recombinant anti-PD-1 monoclonal antibody.
  Arms: Carboplatin /Cisplatin + etoposide + Tislelizumab

SUMMARY:
This is a randomized, controlled, open-label, multicenter clinical study to evaluate the efficacy and safety of carboplatin/cisplatin + etoposide + benmelstobart sequential benmelstobart combined with anlotinib versus carboplatin/cisplatin + etoposide + Tislelizumab sequential Tislelizumab in the first-line treatment of extensive stage small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* The subjects voluntarily joined the study, signed the informed consent, and had good compliance;
* 18 years old ≤age≤ 75 years old (calculated on the date of signing the informed consent);
* Eastern Cooperative Oncology Group (ECOG) score 0 ~ 1;
* Expected survival greater than 12 weeks.
* Histologically or cytologically confirmed Extensive stage small cell lung cancer (ES-SCLC) (according to the Veterans Administration Lung Cancer Society (VALG) disease staging system).
* had not received systemic therapy for ES-SCLC (including systemic chemotherapy, molecular targeted drug therapy, biological therapy and other investigational therapeutic drugs, etc.) or immune checkpoint inhibitor therapy.
* Patients receiving chemoradiotherapy for previously limited-stage SCLC must be treated for cure, and there must be a treatment-free interval of at least 6 months from the last course of chemotherapy, radiotherapy, or chemoradiotherapy to the diagnosis of extensive SCLC.
* Confirmed presence of at least one measurable lesion according to RECIST 1.1 criteria. Note: Measurable target lesions cannot be selected from previous radiotherapy sites. If the target lesion of the previous radiotherapy site is the only alternative target lesion, the investigator should provide pre - and post-imaging data showing significant progression of the lesion.
* Laboratory inspection meets the following standards:

  1. Hemoglobin (HGB) ≥ 90g/L;
  2. Neutrophil absolute value (NEUT) ≥ 1.5× 10 9 /L;
  3. Platelet count (PLT) ≥ 90× 10 9 /L;
  4. Total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal value (ULN);
  5. Alanine transferase (ALT) and aspartate transferase (AST) ≤ 2.5×ULN. ALT and AST≤ 5×ULN if accompanied by liver metastasis;
  6. Serum creatinine (CR) ≤ 1.5×ULN or creatinine clearance (CCR) ≥60 mL /min;
  7. Prothrombin time (PT), activated partial thromboplastin time (APTT), International standardized ratio (INR) ≤ 1.5×ULN (no anticoagulant therapy).
* Women of reproductive age should agree that effective contraception must be used during the study period and for 6 months after the end of the study, and that serum or urine pregnancy tests are negative within 7 days prior to study enrollment; Men should agree that effective birth control must be used during the study period and for 6 months after the end of the study period.

Exclusion Criteria:

* Had or was currently suffering from other malignant tumors within 3 years prior to the first medication. The following two conditions can be included: other malignancies treated with a single operation, achieving continuous 5-year disease-free survival (DFS); Cured cervical carcinoma in situ, non-melanoma skin cancer and superficial bladder tumors [Ta(non-invasive tumor), Tis (cancer in situ) and T1 (tumor infiltrating basal membrane)].
* The presence of diseases affecting intravenous administration, intravenous blood collection, or multiple factors affecting oral medication (such as inability to swallow, chronic diarrhea, and intestinal obstruction);
* The adverse effects of previous treatment did not return to The Common Terminology Criteria for Adverse Events (CTCAE) v5.0 score ≤ 1, except for grade 2 alopecia, grade 2 peripheral neurotoxicity, grade 2 anemia, non-clinically significant and asymptomatic laboratory abnormalities, stable hypothyroidism after hormone replacement therapy and other toxicities deemed by the investigators to be of no safety risk.
* Those who have received major surgical treatment, significant traumatic injury, or major surgery during the intended study treatment period (other than protocol-specified surgery) within the 4 weeks prior to initial medication, or have sustained unhealed wounds or fractures. (Major surgery is defined as surgery at grade 3 and above in the National Surgical Grading Directory 2022 edition).
* Subjects with any bleeding or bleeding event ≥ CTC AE grade 3 within 4 weeks prior to initial dosing.
* Patients who experienced a hyperarterial/venous thrombosis event, such as cerebrovascular accident (including transient ischemic attack), deep vein thrombosis and pulmonary embolism, within 6 months before the first administration of the drug.
* Active viral hepatitis and poorly controlled. Those who meet the following requirements can be screened: HBsAg positive subjects must meet Hepatitis B virus (HBV) DNA quantification <2000 IU/ml (or 1*104 copy/ml) or receive anti-HBV therapy with a 10-fold (1 log) or greater reduction in viral index for at least 1 week prior to study initiation, and subjects are willing to receive anti-HBV therapy throughout the study period; HCV infected persons (HCV Ab or HCV RNA positive) : The investigators judged to be in a stable state or were receiving antiviral therapy at enrollment and continued to receive approved antiviral therapy in the study.
* Patients with active syphilis who need treatment;
* There is a history of active pulmonary tuberculosis, idiopathic pulmonary fibrosis, institutional pneumonia, drug-induced pneumonia, radiation pneumonia requiring treatment, or active pneumonia with clinical symptoms.
* Those who have a history of psychotropic drug abuse and cannot quit or have mental disorders.
* People who are preparing for or have previously received allogeneic bone marrow transplantation or solid organ transplantation.
* History of hepatic encephalopathy.
* Major cardiovascular disease, including any of the following:

  1. According to the New York Heart Association (NYHA) standards of grade II or higher cardiac insufficiency or heart color ultrasound: left ventricular ejection fraction (LVEF) <50%;
  2. There is a history of clinically significant ventricular arrhythmias (such as persistent ventricular tachycardia, ventricular fibrillation, tip torsion ventricular tachycardia) or arrhythmias requiring continuous antiarrhythmic drug treatment;
  3. Unstable angina;
  4. Myocardial infarction occurred within 12 months;
  5. Fridericia- modified QT interval (QTcF) > 450 ms (msec) for men and >470 msec for women (if QTc is abnormal, it can be tested three times at intervals of more than 2 minutes, and its average value is taken);
  6. Congenital long QT syndrome history or family history;
  7. A history of deep vein thrombosis, pulmonary embolism, or any other severe thromboembolism within the 3 months prior to randomization (implantable venous port or catheter-derived thrombosis, or superficial venous thrombosis is not considered "severe" thromboembolism);
  8. Currently receiving or having recently received (within 7 days before the start of study treatment) aspirin (>325mg/ day (maximum antiplatelet dose) or dipyridamole, ticlopidine, clopidogrel, and cilostazol.
* Active or uncontrolled severe infection (≥CTC AE grade 2 infection);
* Patients with renal failure requiring hemodialysis or peritoneal dialysis;
* Have a history of immunodeficiency, including HIV positive or other acquired or congenital immunodeficiency diseases;
* Subjects who require immunosuppressive, systemic, or absorbable topical hormone therapy for immunosuppressive purposes and who continue to use it for 7 days prior to initial administration (except for corticosteroids < 10 mg daily prednisone or other therapeutic hormones);
* People who have epilepsy and need treatment.
* Tumor-related symptoms and treatment:

  1. For subjects who have received chemotherapy, immunotherapy within 3 weeks before the first dose, radiation therapy or small molecule targeted drugs within 2 weeks, or who are still within the 5 half-lives of the drug (as the shortest time of occurrence), the washout period is calculated from the end time of the last treatment;
  2. Within 2 weeks before the first drug use, it has been treated with Chinese patent medicines (including compound Cantharides capsule, Kangai injection, Kanglaite capsule/injection, Aidi injection, Bruceae oil injection/capsule, Xiaoaiping tablet/injection, Cinobufotalin capsule, etc.) with anti-tumor indications specified in the National Medical Products Administration (NMPA) approved drug instructions;
  3. Imaging (CT or MRI) shows that the tumor has invaded important blood vessels, or the investigator determines that the tumor is highly likely to invade important blood vessels during the follow-up study period and cause fatal massive bleeding;
  4. Uncontrolled pleural effusion, pericardial effusion or moderate to severe ascites that still require repeated drainage (investigators' judgment);
  5. Patients with active central nervous system (CNS) metastases and/or cancerous meningitis identified by known or screening tests. Subjects with asymptomatic brain metastases (i.e., no progressive central nervous system symptoms caused by brain metastases, no need for corticosteroids, and the lesion size ≤1.5cm) can participate, but require regular brain imaging as a disease site. (2) Treated subjects with BMS who had stable BMS for at least 2 months (as determined by two imaging studies at least 4 weeks apart after BMS), no evidence of new or expanded BMS, and steroid discontinuation 3 days before study drug administration. Stable brain metastases in this definition should be determined before the first administration of the investigational drug.
  6. Spinal cord compression that was not treated radically by surgery and/or radiotherapy, or previously diagnosed spinal cord compression with no clinical evidence of disease stabilization ≥1 week after treatment prior to randomization.
* Known allergy to study drug excipients, known severe allergic reaction to any monoclonal antibody, history of carboplatin, cisplatin, or etoposide allergy.
* Subjects had previously been treated with other antibodies/drugs targeting immune checkpoints, such as PD-1, PD-L1, CTLA4, etc.
* Previously received treatment with anti-angiogenic drugs such as Anlotinib, Apatinib, and Bevacizumab.
* Participants who had participated in and used other anti-tumor clinical trials within 4 weeks before the first medication.
* In the judgment of the investigator, there is a situation that seriously endangers the safety of the subject or affects the completion of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | From enrollment until the first onset of disease progression or death from any cause, evaluation is expected to take 2 years
  The time from enrollment until the first onset of disease progression or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
12/24 month PFS rate | 12-month, 24-month
  The percentage of subjects with no progression from the first dose to 12 and 24 months of total subjects.
12/24 month Overall survival (OS) rate | 12-month, 24-month
  The number of surviving subjects as a percentage of the total number of subjects from the first dose to 12 and 24 months.
Overall survival (OS) | From randomization to death from all causes, evaluation is expected to take 5 years
  The time between randomization and death from all causes.
Objective response rate (ORR) | Complete response time was achieved, evaluation is expected to take 2 years
  The proportion of subjects achieving complete response (CR) or partial response (PR) was assessed.
Disease Control Rate (DCR) | Complete response time was achieved, evaluation is expected to take 2 years
  The proportion of subjects who achieved complete response (CR), partial response (PR), or stable disease (SD) was assessed.
Incidence of adverse events (AE) and serious adverse events (SAE) | Time of adverse event, evaluation is expected to take 2 years
  The incidence and severity of adverse events were determined according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) v5.0 rating scale.
Patient-reported Outcomes (PRO): Treatment of Cancer Quality of Life Questionnaire - Core 30 | PRO assessments were performed during the screening period, at the end of each even-numbered cycle, at the end of study treatment, and at safety follow-up in the order shown, baseline to 2 years
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 (EORTC QLQ-C30).
  Treatment of Cancer Quality of Life Questionnaire - Core 30 were used to evaluate PRO.
  The EORTC QLQ-C30 v3 questionnaire is an established measure of health-related quality of life (HRQoL)Methods, it is often used as the end point of tumor clinical trials.A score of 0-100, where higher scores indicate greater function, higher HRQoL, or higher symptom levels.
Patient-reported Outcomes (PRO): EORTC QLQ-LC13 | PRO assessments were performed during the screening period, at the end of each even-numbered cycle, at the end of study treatment, and at safety follow-up in the order shown, baseline to 2 years
  EORTC Quality of Life Questionnaire-Lung Cancer 13 (QLQ-LC13) QLQ-LC13 were used to evaluate PRO.The QLQ-LC13 is a 13-item self-filling questionnaire for lung cancer disease that will be associated with the EORTC Use QLQ-C30 together.4-point scale: "Not at all", "somewhat", "quite a bit" and "to a great extent"
Patient-reported Outcomes (PRO): European Quality of Life-5 Dimensions 5 Levels | PRO assessments were performed during the screening period, at the end of each even-numbered cycle, at the end of study treatment, and at safety follow-up in the order shown, baseline to 2 years
  European Quality of Life-5 Dimensions 5 Levels were used to evaluate PRO. EuroQol- 5 Dimension (EQ-5D) is a standardized health status indicator developed by the EuroQol group, which asseses five dimensions: mobility, self-care, general activity, pain/discomfort, and anxiety/depression.Each dimension has five response options that reflect increased difficulty (no problem, some problem, moderate problem, severe)Serious problem (extremely serious problem).

CONTACTS AND LOCATIONS:
Locations (28):
- China (28):
  - Maanshan People's Hospital, Maanshan, Anhui
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Peking University People´s Hospital, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Fujian Medical University 2nd Affiliated Hospital, Quanzhou, Fujian
  - The Second Hospitai. & Clinicae Medical School . Lanzhou University, Lanzhou, Gansu
  - Cancer Hospital of Shantou University Medical College, Shantou, Guangdong
  - Nanfang Hospital, Guangzhou, Guangzhou
  - The fourth hospital of hebei medical university, Shijiazhuang, Hebei
  - Tangshan People's Hospital, Tangshan, Hebei
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Henan Provincial People'S Hospital, Zhengzhou, Henan
  - Henan Cancer Hospital Affiliated Cancer Hospital of Zhengzhou University, Zhengzhou, Henan
  - Huazhong University of Science and Technology Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Baotou Cancer Hospital, Baotou, Inner Mongolia
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - The First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - The First Affiliated Hospital of Shandong First Medical University, Jinnan, Shandong
  - Linyi City People's Hospital, Linyi, Shandong
  - The Second Affiliated Hospital Of Xi'an Jiaotong University, Xi'an, Shannxi
  - Shanxi Cancer hospital, Taiyuan, Shanxi
  - Sichuan cancer hospital, Chengdu, Sichuan
  - Dongyang Municipal People's Hospital, Dongyang, Zhejiang
  - Ningbo Medical Center Lihuili Hospital, Ningbo, Zhejiang
  - Ningbo No.2 Hospital, Ningbo, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang